CLINICAL TRIAL: NCT02652702
Title: Randomized Clinical Trial Comparing the Safety and Efficiency of Circular Stapler-assisted Colostomy With Hand-stitching Colostomy for Colorectal Cancer Patients
Brief Title: Study Comparing Circular Stapler-assisted Colostomy vs Hand-stitching Colostomy of Colorectal Cancer Patients
Acronym: STAPLER
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Not enough patients recruited
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Ding Ke-Feng, Principal Investigator, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRCCZ-D01
Record Dates: First submitted 2015-12-29; First posted 2016-01-12 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Colorectal Carcinoma
Keywords: circular stapler-assisted colostomy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Circular Stapler-assisted Colostomy (Experimental): Using Circular Stapler-assisted Technique to Finish Colostomy after colorectal carcinoma surgery when patient need permanent sigmoid stoma.
  Interventions: Procedure: circular stapler-assisted colostomy
- Hand-stitching Colostomy (Experimental): Using Conventional Hand-stitching Technique to Finish Colostomy after colorectal carcinoma surgery when patient need permanent sigmoid stoma.
  Interventions: Procedure: conventional hand-stitching colostomy

INTERVENTIONS:
Procedure: circular stapler-assisted colostomy — procedure:circular stapler-assisted colostomy device:circular stapler
  Arms: Circular Stapler-assisted Colostomy
Procedure: conventional hand-stitching colostomy — procedure:hand-stitching colostomy
  Arms: Hand-stitching Colostomy

SUMMARY:
Conventional hand-stitching colostomy involves extensive hand-stitching by the surgeon. There are significant variations in the outcome of surgery due to differences in the suture techniques of surgeons. The use of a circular stapler in colostomy seems more rapid and efficient colostomy than the conventional methods.But all those reports are single center retrospective cohort study，no randomized controlled trials have been carried out so far.The aim of this study is to comparing the safety and efficiency of circular stapler-assisted colostomy with conventional hand-stitching colostomy in patients with colorectal carcinoma.

DETAILED DESCRIPTION:
It has been difficult to standardize the pull-out of the colon and the size, shape and sutures of the colostomy due to the different techniques employed and varying levels of skill of surgeons in different regions.Thus, various postoperative colostomy complications are inevitable after surgery. Surgeons have been looking for a simple and efficient way to standardize colostomy and reduce its complications.

So we want to compare the safety and efficiency of circular stapler-assisted colostomy with conventional hand-stitching colostomy in colorectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Receiving permanent colostomy because of colorectal cancer
* Age of ≥18 and ≤80

Exclusion Criteria:

* Not willing or incapable to comply with all study visits and assessments
* Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that puts the patient at high risk for treatment-related complications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
colostomy associated complications | 2 year
  measure the colostomy associated complications,such like hemorrhage,necrosis, stenosis, prolapse, and para-stomal hernia.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital Zhejiang University College of Medicine, Hangzhou, Zhejiang, China